CLINICAL TRIAL: NCT04393454
Title: Phase II Study to Evaluate the Efficacy and Safety of Sirolimus in Subjects With Metastatic, Mismatch Repair Deficient Solid Tumors After Immunotherapy
Brief Title: Study to Evaluate the Efficacy and Safety of Sirolimus in Subjects With Metastatic, Mismatch Repair Deficient Solid Tumors After Immunotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following discussion with the Cancer Center the PI elected to terminate the study.
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10724
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-06

CONDITIONS: Metastatic dMMR Solid Cancer; Solid Tumor; Cancer; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Sirolimus; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sirolimus (Experimental): Participants will be instructed to take 2 milligrams (mg) every day for 28 days (1 cycle). They will be evaluated in the oncology clinic every 2 weeks to make sure they are tolerating the medication well.
  Interventions: Drug: Sirolimus 2mg Tablet

INTERVENTIONS:
Drug: Sirolimus 2mg Tablet — Sirolimus (oral) will be started at 2 mg daily. Sirolimus dosing will be titrated to meet serum trough levels of >8 ng/ml, assayed at 7 days after starting a new dose, by chromatography/mass spectrometry. Once adequate serum levels are met (≥8 ng/ml), the same dosing will be continued until progression of disease as evidenced by imaging, or unacceptable toxicity.

SUMMARY:
To evaluate the efficacy of sirolimus by estimating the overall response rate (ORR) as assessed by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1) in patients with metastatic dMMR solid cancer after immunotherapy (either due to disease progression or to inability to tolerate treatment).

DETAILED DESCRIPTION:
Despite recent therapeutic strategies, including immunotherapy, treatment alternatives for patients with metastatic mismatch-repair deficient (dMMR) solid tumors remain scarce. Pre-clinical data suggests that dMMR tumors are susceptible to rapamycin (sirolimus), an mTOR inhibitor. In these tumors, characterized by higher levels of oxidative stress, sirolimus can exert a cytotoxic effect, led by the failure to repair DNA damage by inhibition of antioxidant enzymes such as FOXO3a triggered by Akt hyperactivation.

This proposal presents a phase 2 clinical trial designed to evaluate the efficacy of sirolimus in patients with dMMR solid tumors after immunotherapy. The investigators hypothesize that sirolimus will increase the overall response rate (ORR) by 20%.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic solid cancer tumor after immunotherapy (either due to progression of disease or inability to tolerate treatment)
* dMMR by immunohistochemistry (IHC) defined as the loss of expression in any of the four major MMR proteins (MLH1, MSH2, MSH6 and PMS2) or by next- generation sequencing (NGS)
* Age older than 18 at the time of informed consent
* Eastern Cooperative Oncology Group performance status of 0-2
* ≥1 measurable lesion based on RECIST, version 1.1 (16)
* Absolute neutrophil count (ANC) ≥1,500 mm3
* Platelet count ≥75,000 mm3
* Hemoglobin ≥ 9 g/dl
* Aspartate aminotransferase (AST) ≤3.0 times the upper normal limit (UNL)
* Alanine aminotransferase (ALT) ≤3.0 times the upper normal limit (UNL) Bilirubin ≤1.5 times the UNL
* Serum creatinine ≤1.5 times the UNL

Exclusion Criteria:

* Received immunotherapy in the prior 21 days.
* Have not recovered from toxicities of prior treatments to at least grade 1.
* Symptomatic central nervous system (CNS) metastases
* Pregnancy or Breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaoyuan Kuang, MD, PhD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled into the study from 11/16/2020 through 12/22/2021 at the Montefiore-Einstein Cancer Center.
Groups:
- Sirolimus: Participants will be instructed to take 2 mg every day for 28 days (1 cycle). They will be evaluated in the oncology clinic every 2 weeks to make sure they are tolerating the medication well.
  Sirolimus 2 milligram (mg) tablet: Sirolimus (oral) will be started at 2 mg daily. Sirolimus dosing will be titrated to meet serum trough levels of >8 ng/ml, assayed at 7 days after starting a new dose, by chromatography/mass spectrometry. Once adequate serum levels are met (≥8 ng/ml), the same dosing will be continued until progression of disease as evidenced by imaging, or unacceptable toxicity.
Period: Overall Study
Arm/Group | Sirolimus
Started | 6
Completed | 4
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: 6 baseline participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: To evaluate the efficacy of sirolimus in patients with metastatic mismatch repair deficient (dMMR) solid cancer after immunotherapy (either due to disease progression or to inability to tolerate treatment), ORR will be determined. For this study ORR will be defined as the percentage of patients who achieve either a complete response (CR = disappearance of all target tumors); or a partial response (PR = ≥30% decrease in the sum of the longest diameters of target tumors) based on Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1) following review of imaging (CT-CAP or PET-CT) data.
Time Frame: Up to approximately 24 weeks after achieving therapeutic sirolimus levels, up to 7 months total
Population: One patient had Stable Disease (SD), but was unable to be analyzed for ORR due to being clinical 'Progression of Disease' (POD) on study. Patient stopped study treatment due to toxicity. As such, only 5 patients were able to evaluated for ORR.
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Participants | 1

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS, the duration of time from treatment initiation to progression of known metastases or new metastatic site, or death from any cause after a timeframe of 24 weeks, will be determined following treatment with sirolimus in patients with metastatic mismatch repair deficient (dMMR) solid cancer after immunotherapy (either due to disease progression or to inability to tolerate treatment). Group median number of months will be reported.
Time Frame: Approximately 24 weeks after sirolimus initiation, up to approximately 7 months total
Population: Progression-free Survival (PFS) was unable to be assessed in 2 of the enrolled patients.
Measure: Median (Full Range); unit: months
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
months | 3.5 [3.3 to 6.0]

3. Secondary Outcome: Response Duration (RD)
Description: RD, defined as the duration of time from documentation of tumor response until the time of disease progression will be determined following treatment with sirolimus in patients with metastatic mismatch repair deficient (dMMR) solid cancer after immunotherapy (either due to disease progression or to inability to tolerate treatment). Group median number of months will be reported.
Time Frame: Up to ~24 weeks from the time of tumor response, up to 7 months total
Population: Response duration was only able to be evaluated in the one patient who showed a Partial Response
Measure: Median (Full Range); unit: months
Arm/Group | Sirolimus
Number analyzed (Participants) | 1
months | 6.0 [6.0 to 6.0]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival, the duration of time from the start of treatment initiation for patients diagnosed with metastatic mismatch repair deficient (dMMR) solid cancer after immunotherapy (either due to disease progression or inability to tolerate treatment) to death from any cause, will be determined. Group median number of months will be reported.
Time Frame: Approximately 24 weeks after sirolimus initiation, up to approximately 7 months total
Population: 2 patients were unable to be evaluated for OS.
Measure: Median (Full Range); unit: months
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
months | 6.1 [3.7 to 6.9]

5. Post Hoc Outcome: Best Overall Response (OR)
Description: To evaluate the efficacy of sirolimus in patients with metastatic mismatch repair deficient (dMMR) solid cancer after immunotherapy (either due to disease progression or to inability to tolerate treatment), the best OR will be determined based on RECIST criteria following review of imaging (CT-CAP or PET-CT) data. Tumor responses will be categorized based on RECIST v1.1 criteria as follows:
  Complete Response (CR): disappearance of all target tumors Partial Response (PR): ≥30% decrease in the sum of the longest diameters of target tumors Progressive Disease (PD): at least 20% increase in sum of diameters of target tumor (noting smallest sum on study); absolute increase of 5mm must be demonstrated Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD Inevaluable/Not Evaluable (NE): No imaging taken/no measurement performed
Time Frame: Up to approximately 24 weeks after achieving therapeutic sirolimus levels, up to 7 months total
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 6
Participants
  CR | 0
  PR | 1
  SD | 3
  PD | 1
  NE | 1

ADVERSE EVENTS:
Time Frame: Approximately 24 weeks following initiation of treatment, up to 7 months total.
Arm/Group | Sirolimus
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=6)
Abdominal Pain (Gastrointestinal disorders) | 1 — Hospitalized, Grade 3
Vomiting (Gastrointestinal disorders) | 1 — Hospitalized, Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=6)
Fatigue (General disorders) | 3 — All Grade 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 — Verbatim Term: Hoarse Voice. Grade 1
Anorexia (Metabolism and nutrition disorders) | 2 — Grade 1
Neuropathy (Nervous system disorders) | 1 — Verbatim Term. Grade 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 — One with intermittent back pain. Other with left, lateral back pain. Other unspecified. All Grade 1
Abdominal Pain (Gastrointestinal disorders) | 1 — Intermittent. Grade 1
Dysuria (Renal and urinary disorders) | 1 — Grade 1
Diarrhea (Gastrointestinal disorders) | 3 — 1 intermittent. All Grade 1
Hypertension (Cardiac disorders) | 1 — Grade 3
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 2 — Both Grade 1
Mucositis, Oral (Gastrointestinal disorders) | 1 — Grade 1
Acute Kidney Injury (Renal and urinary disorders) | 1 — Grade 1
Headaches (Nervous system disorders) | 1 — Intermittent, Grade 1
Weight Loss (Investigations) | 1 — Grade 1
Pain (Musculoskeletal and connective tissue disorders) | 1 — Verbatim Term: Knee Pain
Edema Limbs (General disorders) | 2 — Verbatim Term: Bilateral, Lower Extremity Edema
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 1
Hypokalemia (Metabolism and nutrition disorders) | 1 — Grade 1
Urinary Tract Infection (Infections and infestations) | 1 — Grade 1
COVID Infection (Infections and infestations) | 1 — Verbatim Term. Grade 1
Anemia (Blood and lymphatic system disorders) | 2 — Both Grade 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT04393454/Prot_SAP_000.pdf